CLINICAL TRIAL: NCT05702138
Title: Improving Balance and Mobility After Traumatic Brain Injury: A Randomized Controlled Trial Evaluating High Intensity Step Training
Brief Title: High Intensity Step Training After Traumatic Brain Injury
Acronym: B-HIST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Craig Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB#1947316-1
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Traumatic Brain Injury
Keywords: balance; mobility; physical therapy
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Gait and Balance Training (CGBT) (Active Comparator): The current approach for walking retraining, Conventional Gait and Balance Training (CGBT) focuses on walking training in a variety of conditions, obstacle management training, functional independence training, strength training, and standing dynamic balance training.
  Interventions: Other: Physical therapy
- High Intensity Step Training (HIST) (Experimental): High Intensity Step Training (HIST) focuses on the repetition of stepping at higher cardiovascular intensities and yielding a greater number of steps per training session.
  Interventions: Other: Physical therapy
- High Intensity Step Training with Virtual Reality (HISTVR) (Experimental): The third arm combines virtual reality with HIST, designed to increase cortical excitability while concurrently activating the neuromuscular system.
  Interventions: Other: Physical therapy

INTERVENTIONS:
Other: Physical therapy — The study evaluates three physical therapeutic approaches to improve mobility and balance after traumatic brain injury (TBI).

SUMMARY:
This study will explore whether the types and intensity of the interventions being delivered will yield measurable cognitive benefits in addition to improved mobility and balance.

The study evaluates three therapeutic approaches to improve mobility and balance after traumatic brain injury (TBI): Conventional Gait and Balance Training, high intensity step training, and high intensity step training with virtual reality.

DETAILED DESCRIPTION:
Individuals with traumatic brain injury (TBI) walk more slowly, demonstrate greater imbalance, and have reduced endurance. There is strong evidence that a single bout of physical activity has substantial cognitive benefits among older adults and stroke survivors, yet similar studies have not been conducted in TBI. This study will explore whether the types and intensity of the interventions being delivered will yield measurable cognitive benefits in addition to improved mobility and balance.

The study evaluates three therapeutic approaches to improve mobility and balance after TBI: the first approach, Conventional Gait and Balance Training (CGBT), represents the current approach for walking retraining. CGBT focuses on walking training in a variety of conditions, obstacle management training, functional independence training, strength training, and standing dynamic balance training. The second approach, high intensity step training (HIST), focuses on the repetition of stepping at higher cardiovascular intensities and yielding a greater number of steps per training session with promising evidence already published in stroke and spinal cord injury (SCI). The third approach combines virtual reality with HIST, designed to increase cortical excitability while concurrently activating the neuromuscular system.

ELIGIBILITY:
Inclusion Criteria:

* TBI definition: damage to brain tissue caused by an external mechanical force as evidenced by loss of consciousness (LOC) or post traumatic amnesia (PTA) due to brain trauma or by objective neurological findings that can be reasonably attributed to TBI on physical examination or mental status examination
* Less than 6 months post injury at time of consent
* Weight less than 298 pounds and height less than 6'2" (based on treadmill contraindications)
* Intact skin (no open lesions/bandages) in the area of treadmill harness contact
* Able to walk ten feet requiring the physical assistance of not more than two people and/or bracing, assistive devices
* Impaired walking speed of < than 1.4 meters/second
* Ability to follow directions/standardized instructions
* Minimum 18 years of age at consent
* Completing or have completed initial inpatient rehabilitation for TBI
* O-Log score of at least 20
* Medically cleared for HIST by a physician

Exclusion Criteria:

* Uncontrolled cardiopulmonary, metabolic, or infectious disorder
* History of orthopedic or additional neurological disorder that limited motor function before TBI
* Any reason that, in the opinion of the study investigators or medical team, would interfere with completing the study protocol such as behavioral concerns
* Uncontrolled seizure disorder
* Pregnant or lactating females
* Current participation in any other interventional trials
* History of an untreated or a poorly controlled psychiatric condition such as depression, schizophrenia, or bipolar disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Walking Speed | 6 Weeks
  10 Meter Walk Test (10MWT)

SECONDARY OUTCOMES:
Walking Endurance | 6 Weeks
  6 Minute Walk Test (6MWT)
Balance | 6 Weeks
  Functional Gait Assessment and Berg Balance Scale (FGA) and (BBS)
Participant Enjoyment | 6 Weeks
  Physical Activity Enjoyment Scale

OTHER OUTCOMES:
Cognition | 6 Weeks
  Brief Test of Adult Cognition by Telephone (BTACT):

CONTACTS AND LOCATIONS:
Overall Officials: Candy Tefertiller, DPT, PhD, Principal Investigator — Craig Hospital
Locations (1):
- Craig Hospital, Englewood, Colorado, United States